CLINICAL TRIAL: NCT04169867
Title: Polish Microbiome Map
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ardigen (Industry)
Collaborators: The Institute of Bioorganic Chemistry, Polish Academy of Sciences (Unknown); National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: MMP; POIR.04.01.02-00-0025/17 (Other Grant/Funding Number: The National Centre for Research and Development)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Melanoma; Healthy Volunteers; Microbiome; Metagenome; Immunotherapy
Keywords: Microbiome; Melanoma; Healthy Volunteers; Immunotherapy; Stool samples; Cancer; Metagenome; Neoplasms; Intestinal microbiota; Nivolumab; Ipilimumab; Atezolizumab
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Nivolumab; Ipilimumab; atezolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: This cohort will consist of 1000 healthy volunteers from Poland.
- Melanoma: This cohort will consist of 160 patients with melanoma.
  Interventions: Biological: Collection of stool samples

INTERVENTIONS:
Biological: Collection of stool samples — Patients receiving routine treatment (immunotherapy using anti-PD1 / anti-PDL1 and / or anti CTLA4 antibodies), financed by the Polish National Health Fund (NFZ).
  Other Names: Nivolumab; Ipilimumab; Atezolizumab
  Groups: Melanoma

SUMMARY:
Knowledge about the correlations between the composition of the gut microbiome and a wide range of diseases has substantially increased in recent years. Nonetheless, there is no reference set of information about the microbiome in Poland. The development of such a reference will allow polish scientists conducting research in the field of interaction between gut flora components and such characteristics as lifestyle, certain diseases or patient's responses for treatment. Following the example of such countries as the United States, investigators propose to build a unique set of scientific processed information describing the variability of the polish population microbiome (Polish Microbiome Map). The investigators will provide a reliable dataset that will characterize the gut microbiomes and their diversity in the polish population. Additionally, thanks to the creation of the standard protocol for microbiome data collection the research conducted by the MMP users will be comparable with the information deposited in MMP.

ELIGIBILITY:
Inclusion Criteria for Healthy Volunteers group:

* Men or women ≥18 years of age
* Patients with informed consent to participate in the study.

Inclusion Criteria for Melanoma group:

* Men or women ≥18 years of age
* Patients with melanoma
* Patients with informed consent to participate in the study.
* Patients receiving routine treatment (immunotherapy using anti-PD1 / anti-PDL1 and / or anti CTLA4 antibodies), financed by the Polish National Health Fund (NFZ).
* The applied immunotherapy should be the first or second line of treatment.

Exclusion Criteria:

* Patients or Healthy Volunteers who are unable to understand, read and / or sign the informed consent
* Patients or Healthy Volunteers who can not collect stools
* Patients with a fecal transplant
* The applied immunotherapy is not the first or second line of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers or oncology patients with primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1160 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbial diversity in stool samples | Inclusion
  Microbial DNA - stool samples sequenced by next-generation sequencing platform.
Eating habits and health survey | Inclusion
  It includes questions about healthy volunteers' and patients' eating habits that may relate to their health.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Philips, PhD, Principal Investigator — The Institute of Bioorganic Chemistry, Polish Academy of Sciences; Jan Majta, Principal Investigator — Ardigen
Locations (1):
- The Institute of Bioorganic Chemistry, Polish Academy of Sciences, Poznan, Poland